CLINICAL TRIAL: NCT04752943
Title: Tips By Text: Using Text Messages to Support Clinic Parents and Improve Child School Readiness Outcomes
Brief Title: Leveraging Clinic to Promote Literacy in Young Children
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Stanford University (Other)
Collaborators: Santa Clara Valley Medical Center (Other)
Responsible Party: Principal Investigator, Lisa Chamberlain, Professor of Pediatrics, Stanford University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 42320
Record Dates: First submitted 2021-02-02; First posted 2021-02-12 (Actual); Last update posted 2021-03-29 (Actual); Status verified 2021-03

CONDITIONS: Literacy
Keywords: school readiness
MeSH Terms: conditions — Literacy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Children and caregivers receiving TipsByText messages (Experimental)
  Interventions: Other: Tips By Text Messages
- Children and caregivers not receiving TipsByText texts (No Intervention)

INTERVENTIONS:
Other: Tips By Text Messages — Texts sent to caregivers meant to increase parent child interaction around literacy, sent to participants 3 x a week for 7 months
  Arms: Children and caregivers receiving TipsByText messages

SUMMARY:
Our primary aim of this study is to assess the impact of an early literacy text messaging program (TipsByText, TbT) for parents of children between 3 to 4-years old during an office visit without access to preschool. To assess this aim, our objectives are to specifically assess (1) child literacy using the Phonological Awareness Literacy Screening Tool (PALS-PreK) and (2) caregiver involvement using the Parent Child Interactivity Scale (PCI) pre- and post-intervention, comparing with a control group not receiving the TipsByText intervention. A secondary outcome of this study is to compare trust among families that participate in the Tips by Text (TbT) Program with families that do not participate in TbT using the Trust Evaluation Scale. Children will complete the PALS-PreK and caregivers of the children will complete the PCI and Trust Evaluation Scales.

ELIGIBILITY:
Inclusion Criteria:

* Parents of participants must be last least 18 years of age.
* Parents must be English and Spanish speaking, as the Tips by Text texting platform is currently in those languages.
* Child must be 3-5 years old at the time of their clinic visit.

Exclusion Criteria:

* Parent does not speak English or Spanish. This applies given that the texting intervention has the capacity to be conducted in these two languages.
* Parent does not have cell phone that would allow texting.
* For the literacy texting intervention, the child must NOT be enrolled in Head Start,Transitional Kindergarten or other subsidized preschool. Parents will be provided with a list of preschools that would warrant exclusion. Childcare is ok. For the trust and no-show evaluation arm, participants may be enrolled in any form of early childhood education.
* Child is currently receiving services for delay (speech, motor, or cognitive). If the child briefly received services for delays over a year before start date of the study, they are still eligible.

Ages: 3 Years to 5 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 381 (Actual)
Dates: Start 2017-10-16 (Actual); Primary Completion 2019-07-26 (Actual); Study Completion 2019-07-26 (Actual)

PRIMARY OUTCOMES:
Change in child literacy measured by the Phonological Awareness Literacy Screening Tool (PALS-PreK) Score | Baseline and month 9
  The PALS-PreK measures preschoolers' knowledge of literacy fundamentals: name writing, alphabet knowledge, sound awareness, print and word awareness, rhyme awareness, and nursery rhyme awareness. The English and Spanish PALS-PreK versions slightly differ in content, thus we standardized composite scores for both the pre and post score by language to allow fair comparisons. Lower-case alphabet recognition or letter sounds was not included in the total score for English or Spanish. Score range for English was 0 to 73 and for Spanish was 0 to 94, with higher score indicating better outcome
Change in caregiver involvement measured by the Parent Child Interactivity Scale (PCI) | Baseline and month 9
  The Parent Child Interactivity Scale (PCI) uses parent self-assessment and a four-point Likert scale for five items assessing reading, such as "Looked at pictures together in a book", and ten items assessing other literacy activities, such as "Practiced rhyming words". We calculated scores for reading (PCI Read), for other activities (PCI Activities), and a composite score was calculated (PCI Total). Items ranged from 0 to 3 for 15 items, thus score ranged from 0 to 45, with higher score indicating better outcome.

SECONDARY OUTCOMES:
Change in parent trust in pediatricians using Wake Forest Physician Trust Scale | Baseline and month 9
  Physician trust is measured by the sum of the 10 item scores (reverse-scored for negative items), ranging from 10 to 50, with a higher score indicating more trust.

CONTACTS AND LOCATIONS:
Overall Officials: Lisa J Chamberlain, MD, MPH, Principal Investigator — Stanford University; Janine Bruce, MPH, DrPH, Study Director — Stanford University; Susanna Loeb, PhD, Study Director — Brown University
Locations (1):
- Valley Medical Center, San Jose, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Doss C, Fahle EM, Loeb S, York BN. More Than Just a Nudge Supporting Kindergarten Parents with Differentiated and Personalized Text Messages. Journal of Human Resources. 2019;54(3):567-603
- [Background] Invernizzi M, Sullivan A, Meier J, Swank L. Phonological awareness literacy screening (PALS) PreK. . Richmond, VA: University of Virginia. 2004.
- [Background] York BN, Loeb, S., & Doss, C. One Step at a Time: The Effects of an Early Literacy Text-Messaging Program for Parents of Preschoolers Journal of Human Resources 54(3), 537-566. 2019.
- [Derived] Chamberlain LJ, Bruce J, De La Cruz M, Huffman L, Steinberg JR, Bruguera R, Peterson JW, Gardner RM, He Z, Ordaz Y, Connelly E, Loeb S. A Text-Based Intervention to Promote Literacy: An RCT. Pediatrics. 2021 Oct;148(4):e2020049648. doi: 10.1542/peds.2020-049648. Epub 2021 Sep 20. PMID 34544847